CLINICAL TRIAL: NCT03540212
Title: Clinical Pharmacokinetics, Safety and Efficacy Study of Daclatasvir/Sofosbuvir in Adolescents Aged 12 to 18 Years Old With Hepatitis C Virus: A Preliminary Study
Brief Title: Clinical Pharmacokinetics of Daclatasvir/Sofosbuvir in Adolescents With Hepatitis C Virus
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Manal Hamdy El-Sayed, Professor of Pediatrics, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMASU P69a/2017
Record Dates: First submitted 2018-02-23; First posted 2018-05-30 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Chronic HCV Infection
MeSH Terms: interventions — daclatasvir; Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Daclatasvir and sofosbuvir (Experimental): Daclatasvir and sofosbuvir
  Single arm intervention open label trial for single tablet (Daclatasvir 90 mg and Sofosbuvir 400mg and ) Daclatasvir 90 mg for 12 weeks
  Interventions: Drug: Daclatasvir and sofosbuvir

INTERVENTIONS:
Drug: Daclatasvir and sofosbuvir — Daclatasvir is a DAAs that can inhibit the HCV non-structural (NS) 5A protein when used in combination with other HCV-therapies. It has a linear, non-time-dependent pharmacokinetic profile and nanomolar potency in vitro against HCV genotypes 1-6. It is excreted primarily via faeces, about 88% in an unchanged form while renal excretion accounts for approximately 7% of its elimination.
  DOSE OF SOFOSBUVIR: 400 mg tablet orally once daily with food (in the morning) for 12 weeks for adolescents with liver fibrosis Metavir score F0-F2.
  DOSE OF DACLTASVIR: 60 mg tablet orally once daily with food (in the morning) for 12 weeks for adolescents with liver fibrosis Metavir score F0-F2.
  Other Names: DCV-SOF; Sofosbuvir-Daclatasvir

SUMMARY:
This is an interventional Phase II/III, single center, single arm clinical trial to assess the pharmacokinetics, efficacy, safety and tolerance of daclatasvir plus sofosbuvir in treatment-naïve, non-cirrhotic adolescents with chronic HCV GT-4 infection.

A single-arm evaluation of daclatasvir/sofosbuvir will focus on the pharmacokinetics, efficacy and safety

All enrolled patients will receive daclatasvir 60 mg orally once daily plus sofosbuvir at a dose of 400 mg orally once daily for 12 weeks.

DETAILED DESCRIPTION:
This is an interventional Phase II/III, single center, single arm clinical trial to assess the pharmacokinetics efficacy, safety, and tolerance of daclatasvir plus sofosbuvir in treatment-naïve, non-cirrhotic adolescents with chronic HCV GT-4 infection.

A single-arm evaluation of daclatasvir/sofosbuvir will focus on the efficacy, safety and pharmacokinetics, confirm the favorable pharmacological profile.

All enrolled patients will receive daclatasvir 60 mg orally once daily plus sofosbuvir at a dose of 400 mg orally once daily for 12 weeks.

Patients will be followed closely for disease progression and any hypersensitivity or adverse reactions due to therapy. Laboratory values to be monitored at baseline: Serum creatinine, bilirubin, AST, ALT, HCV viral load (VL).

Fifty patients will be included; the first twenty patients will be candidates for pharmacokinetic assessment. All patients (50), will be candidates for safety and efficacy assessment after verifying the PK results ''phase II''. Patients will be recruited at Ain Shams University hospitals, Egypt. The study will be conducted after approval of the corresponding research ethical committee and obtaining an informed consent from the parents/guardians and an assent from the patients.

Patients will be requested to come for 2 screening visits, at the first day of therapy, weekly during the first four weeks, at the end of week 8 and week 12. Patients who will complete their treatment schedule will be scheduled for a visit after 12 weeks from end of therapy for assessment of sustained virological response (SVR). The total number of visits are 9. Duration of follow up will be 24 weeks from treatment initiation in addition to the screening period (2-4 weeks).

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents (ages 12- 18 years) and/ or weight ≥ 35 kg
2. HCV genotype 4 infected
3. Naïve non-cirrhotic population with FIB Score: F0 to F3.
4. Screening laboratory values within define thresholds
5. Both sex
6. Evidence of HCV infection determined by positive anti-HCV antibody and HCV RNA by polymerase chain reaction (PCR)
7. HCV treatment-naïve
8. Absolute neutrophil count ≥ 1,500/mm3
9. Hemoglobin level ≥ 10 g/dL
10. Platelets > 75000 cells/mm3
11. Albumin > 3.5 mg/dL
12. PT < 3 sec above control and INR within accepted range
13. Random glucose level within normal range
14. Serum creatinine < 1.5 mg/dL
15. Biopsy is not required for study entry.
16. Signing informed consent by parents and patient assent

Exclusion Criteria:

1. Previous treatment for HCV.
2. History of clinically significant illness or any other medical condition that may interfere with individuals' treatment, assessment, or compliance with protocol.
3. Co-infection with HIV, acute hepatitis A virus, or hepatitis B virus
4. Clinical hepatic decompensation (i.e., ascites, encephalopathy or variceal hemorrhage)
5. Pregnant or nursing females
6. Use of any illicit concomitant medications as within 28 days of the Day 1
7. Renal dysfunction
8. Ongoing treatment with Prohibited drugs.
9. Chronic liver disease due to a cause other than HCV e.g. autoimmune disease, Wilson disease,…etc.
10. Alfa-fetoprotein level >50 ng/mL
11. Serum creatinine >1.5 mg/dL
12. Simultaneous acute hepatitis A infection
13. Known hypersensitivity to daclatasvir or sofosbuvir
14. History of gastrointestinal disease or surgical procedure
15. Blood /blood product transfusion within 4 weeks prior to study
16. Systemic corticosteroid use for more than 2 weeks (pulmonary/nasal administration was permitted)
17. Psychiatric hospitalization, suicide attempt or disability resulting from psychiatric illness within the prior 5 years
18. Clinically relevant alcohol or drug abuse within 12 months of screening
19. Ongoing treatment with any medications interacting with daclatasvir/sofosbuvir

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-12-10 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of the pharmacokinetics of DCV-SOF | Blood samples will be collected on day 8 of therapy
  Blood samples (3 mL) will be collected to measure dactalasvir concentrations from pediatric patients using a nine-point plasma schedule (pre-dose, 0.5,1, 2, 4, 8, 12, and 24 h post-dose) on day 8 of therapy.
  (This will be a total of 27 mL/patient, which is well below the maximum allowed internationally recognized value of blood loss is 2.4mL/kg in a 4 month period. Any deviations from nominal sampling times should be recorded.
  AUCtau which is defined as the concentration of drug over time (area under the plasma concentration versus time curve over the dosing interval will be calculated

SECONDARY OUTCOMES:
Measurement of Number of Participants With sustained virological response (SVR12), 12 weeks after discontinuation of therapy with daclatasvir-sofosbuvir (DCV-SOF). | 12 weeks after discontinuation of therapy with daclatasvir-sofosbuvir (DCV-SOF).
  Number of Participants With sustained virological response at 12 Weeks after end of study drug treatment (SVR12) will be recorded, participant will be considered to have achieved SVR12 if HCV RNA is less than the lower limit of quantification of <15 IU/ml) at 12 weeks after the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Manal H El-Sayed, MD, Principal Investigator — Professor of Pediatric, Faculty of Medicine, Ain Shams University, Egypt
Locations (1):
- Pediatric Department, Faculty of Medicine, Ain Shams University, Cairo, Non-US, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al-Nahari MM, Abbassi MM, Ebeid FS, Hassany M, El-Sayed MH, Farid SF. Pharmacokinetics of daclatasvir in Egyptian adolescents with genotype-4 HCV infection. Antivir Ther. 2020;25(2):101-110. doi: 10.3851/IMP3357. PMID 32367815